CLINICAL TRIAL: NCT01329445
Title: Post Market, Longitudinal Data Collection Study of DeNovo NT for Articular Cartilage Defects of the Knee
Brief Title: DeNovo NT Longitudinal Data Collection (LDC) Knee Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zimmer Orthobiologics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSU2010-22B
Record Dates: First submitted 2011-04-01; First posted 2011-04-06 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-12

CONDITIONS: Degenerative Lesion of Articular Cartilage of Knee; Osteochondritis Dissecans
Keywords: Cartilage repair; Articular cartilage defects
MeSH Terms: conditions — Osteochondritis Dissecans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- DeNovo NT patient: Patients who have received or who are scheduled to receive a DeNovo NT graft for repair of 1-2 knee cartilage lesions.
  Interventions: Other: DeNovo NT, Natural Tissue Graft

INTERVENTIONS:
Other: DeNovo NT, Natural Tissue Graft — DeNovo NT Natural Tissue Graft of 1 or 2 lesions up to 5 cm squared in area.
  Other Names: DeNovo NT

SUMMARY:
The purpose of this study is to evaluate the long-term outcomes of DeNovo NT, a tissue product used for the repair of cartilage damage in the knee. This product has been on the market since 2007 and implanted in more than 10,000 patients around the country.

DETAILED DESCRIPTION:
Knee cartilage injury is a major cause of pain and functional impairment in young to middle age adults, and can lead to progressive joint degeneration. Adult cartilage has little regenerative capacity and many of the current treatment options have limited or unknown durability. DeNovo NT is an allogeneic tissue graft, prepared from donated juvenile cartilage, which has been shown to have a higher chondrogenic potential than adult cartilage. The graft involves a single surgery with no need for scaffolds, flaps or donor-site morbidity. This study will follow the long-term outcomes and durability of DeNovo NT in patients grafted with this product in the knee, for up to five years. It will enroll subjects prospectively (at the time of surgery) and retrospectively (those who have been previously implanted). Data will be collected on patient-reported outcomes, results of knee examinations, and reoperations and revisions.

ELIGIBILITY:
Inclusion Criteria:

* Has a contained articular cartilage lesion(s) of the knee or Osteochondritis Dissecans OCD lesion(s) of the knee for which arthroscopic or surgical intervention is warranted, OR Has had prior treatment with DeNovo NT for a contained articulare cartilage lesion(so of the knee or Osteochondritis Dissecans OCD lesion(s) of the knee
* Has voluntarily signed the IRB approved Informed Consent
* Is of stable health and is able to undergo surgery
* Is male or female over the age of 18 years
* Is physically and mentally willing and able to comply with post-operative rehabilitation and routinely scheduled clinical visits

Exclusion Criteria:

* Displays a high surgical risk as determined by the investigative surgeon
* Is pregnant or breast-feeding
* Has a clinically diagnosed autoimmune disease
* Has an active joint infection or history of chronic joint infection at the surgical site
* Has damage to the subchondral bone that has not/will not be repaired prior to DeNovo NT treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being recommended for arthroscopic or surgical intervention for articular cartilage lesionis of the knee
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2011-02; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Mean scores from patient-reported clinical outcome surveys | 5 years

SECONDARY OUTCOMES:
Incidence of reoperations and revision surgeries | 5 Years

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Specialized Orthopaedic Surgery & Spine Center, Huntsville, Alabama
  - Naval Medical Center San Diego, San Diego, California
  - Colorado Orthopedic Consultants, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Midwest Orthopaedics at Rush Univ Hospital, Chicago, Illinois
  - OrthoIndy, Greenwood, Indiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - New Mexico Orthopaedic Associates, Albuquerque, New Mexico
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Specialized Orthopaedics & Sports Medicine, Columbus, Ohio
  - Cleveland Clinic Sports Health Center, Garfield Heights, Ohio
  - University of Virginia, Charlottesville, Virginia
  - Jordan Young Institute, Virginia Beach, Virginia
  - Aurora Baycare Medical Center, Green Bay, Wisconsin
  - Dean Clinic, Madison, Wisconsin